CLINICAL TRIAL: NCT04478955
Title: Effect of Pencil Eyeliners and Waterproof Mascara on Tear Stability Tests and Meibomography
Brief Title: Effect of Eye Make up on Ocular Surface
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Eylül Ercan, Doctor, Erol Olcok Corum Training and Research Hospital
Other Study IDs: Corum State Hospital
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Meibomian Gland Dysfunction
Keywords: meibomian, eyeliner
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Wettability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal: no make up
  Interventions: Diagnostic Test: Schirmer test
- eyeliner only: three days a week at least for 6 months
  Interventions: Diagnostic Test: Schirmer test
- mascara only: three days a week at least for 6 months
  Interventions: Diagnostic Test: Schirmer test
- eyeliner and mascara: three days a week at least for 6 months
  Interventions: Diagnostic Test: Schirmer test

INTERVENTIONS:
Diagnostic Test: Schirmer test — Tear tests Meibomian gland grading test
  Other Names: Non contact tear break up test; Meibomography

SUMMARY:
The aim of this study is to compare the degree of tear film instability and severity of meibomian gland loss between subjects who use eyeliner, mascara, a combination of both and those who do not use eyeliner.

ELIGIBILITY:
Inclusion Criteria:

To use eyeliner/mascara or combined for at least 3 days for 6 months for study groups No routine eye make up use for the cıontrol group

-

Exclusion Criteria:

* any systemic or ocular disease taht can affect ocular surface

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — eye make up use
Study Population: 18 to 35 year old females with eyeliner, mascara or combined use for study groups 18 to 35 year old females with no make up use for control group
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-29 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Schirmer test | 5 minutes
  Tear measurement

SECONDARY OUTCOMES:
Non contact tear break up test | 17 seconds
  tear stability calculation
Meibomography | 2 minutes
  Meibomian gland loss grading

CONTACTS AND LOCATIONS:
Locations (1):
- ErolOlcok Corum WEducatin and Research Hospital, Çorum, Turkey (Türkiye)